CLINICAL TRIAL: NCT05281406
Title: Additional Chemotherapy for EGFRm Patients with the Continued Presence of Plasma CtDNA EGFRm At Week 3 After Start of Osimertinib 1st-line Treatment (PACE-LUNG)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Martin Sebastian, Principal Investigator, Goethe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PACE LUNG
Record Dates: First submitted 2022-02-01; First posted 2022-03-16 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: NSCLC Stage IIIB; NSCLC Stage IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: Phase II prospective non-randomized biomarker-enriched single arm trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Osimertinib in combination with platinum-based chemotherapy (Experimental): all patients received a platinum-based chemotherapy (carboplatin/pemetrexed or cisplatin/pemetrexed) for a maximum of 4 cycles (q3w) in combination with 80 mg Osimertinib daily
  Interventions: Drug: Osimertinib; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Osimertinib — 80 mg daily or reduced dose 40 mg daily
  Other Names: Tagrisso
Drug: Pemetrexed — 500 mg/m² i.v. d1 of every 21-day cycle for a maximum of 4 cycles
Drug: Cisplatin — 75mg/m² i.v. d1 of every 21-day cycle for a maximum of 4 cycles
Drug: Carboplatin — AUC 5 mg/mL/min i.v. d1 of every 21-day cycle for a maximum of 4 cycles

SUMMARY:
PACE is a prospective multicenter single-arm investigator-initiated phase II trial that examines the value of a treatment escalation strategy by the addition of platinum-based doublet chemotherapy to osimertinib in patients with treatment-naïve NSCLC harboring L858R or del19 EGFR mutation who are suspected to have poor response upon single-agent TKI treatment.

DETAILED DESCRIPTION:
Hypothesize, that in patients with on-label osimertinib 1st-line treatment of stage IIIB or IV NSCLC, a biomarker-driven escalation of osimertinib therapy with a platinum-based chemotherapy regimen will effectively enhance PFS and subsequently OS. Lack of EGFRm clearance after an osimertinib treatment period of 3 weeks as assessed by liquid biopsy will be used to predict sub-optimal response. In these patients, treatment will be escalated after approx. 7 weeks of on-label osimertinib monotherapy by adding up to 4 cycles of a combination regimen of pemetrexed and cisplatin or carboplatin. Patients with complete EGFR plasma clearance will continue to receive standard of care osimertinib and will not be eligible for the study. Primary outcome measure will be PFS, which will be compared to historical data on TKI monotherapy from persistent EGFR shedder from the FLAURA trial.

ELIGIBILITY:
Inclusion Criteria:

Pre-Screening Phase

1. Provision of written informed consent for the pre-screening phase.
2. Age ≥ 18 years
3. Histologically confirmed stage IIIB or IV NSCLC
4. Tumor positive for Ex19del or L858R EGFR mutation assessed according to local standard.
5. Planned treatment with osimertinib 80mg/d 1st-line as SoC or ongoing treatment for a maximum of 28 days
6. Available radiographic chest and abdominal CT or MRI scans performed up to 42 days before initial osimertinib treatment
7. Previously untreated with systemic treatment given as primary therapy for advanced or metastatic disease, except for osimertinib for a maximum of 28 days (see above)
8. At least one measurable site of disease as defined by RECISTv1.1 criteria
9. Female subjects of childbearing potential (WOCBP) should be using highly effective contraceptive measures and must have a negative urine or serum pregnancy test within 7 days prior to start of study treatment and must not be breast-feeding prior to start of trial. Further information in Appendix 20.7 (Definition of Women of Childbearing Potential and Acceptable Contraceptive Methods)
10. Non-child-bearing potential must be evidenced by fulfilling one of the following criteria at screening:

    * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
    * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution.
    * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation

Treatment Phase

1. Provision of informed consent for the screening and treatment phase prior to any study specific procedures, including screening evaluations that are not SoC.
2. Persistent mEGFR ctDNA signal 21 to 28 days after osimertinib initiation for advanced of metastatic ex19del or L858R EGFR mutation positive NSCLC as assessed by a liquid biopsy during the pre-screening phase of the trial in the central laboratory.
3. ECOG performance status 0-2.
4. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.
5. Osimertinib no longer than 10 weeks before start of chemotherapy in the treatment phase

Exclusion Criteria:

Pre-Screening Phase

1. History of another primary malignancy. Exceptions are:

   * Malignancy treated with curative intent and with no known active disease ≥6 months before the first dose of IMP, and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease
2. History of leptomeningeal carcinomatosis
3. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study, or during the follow-up period of an interventional study
4. Previous enrolment in the present study.

Treatment Phase

1. Symptomatic CNS metastases. [Patients with asymptomatic brain metastases may be included.]
2. History of leptomeningeal carcinomatosis
3. Currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3 weeks prior) (Appendix 20.5). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
4. Osimertinib had to be withheld or administered at reduced dosage for toxicity management for more than 7 days or persistent unresolved toxicities which preclude study treatment.
5. Any unresolved toxicities other than osimertinib from prior therapy greater than CTCAE grade 1 at the time of starting study treatment, with the exception of alopecia and grade 2 prior platinum-therapy-related neuropathy.
6. History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib. History of hypersensitivity to any of the chemotherapy drugs used.
7. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
8. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
9. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value
   2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block.
   3. Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < LLN; Serum/plasma magnesium < LLN; Serum/plasma calcium < LLN), congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes. [Note: Electrolyte abnormalities (hypokalaemia, hypomagnesaemia, hypocalcaemia) can be corrected to be within normal ranges prior to first dose. No more than two re-tests may be performed in order to meet this criterion.]
10. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
11. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

    1. Absolute neutrophil count below lower limit of normal (<LLN) *
    2. Platelet count below lower limit of normal (<LLN) *
    3. Hemoglobin <90 g/L *

       * The use of granulocyte colony stimulating factor support, platelet transfusion and blood transfusions to meet these criteria is not permitted.
    4. Alanine aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
    5. Aspartate aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases;
    6. Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome [unconjugated hyperbilirubinaemia] or liver metastases;
    7. Serum creatinine >1.5 times ULN concurrent with creatinine clearance <60 mL/min [calculated by Cockcroft and Gault equation]-confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
    8. INR ≤ 1.4 or aPTT ≤ 40 sec during the last 7 days before chemotherapy [Subjects under therapeutic anticoagulation are permitted.]
12. Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
13. Women who are pregnant or breast-feeding
14. Male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 4 months (male patients) or 6 weeks (female patients) after the last dose of osimertinib and 6 months after the last dose of chemotherapy.
15. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].
16. Treatment with an investigational drug within five half-lives of the compound or 3 months, whichever is greater.
17. Any chemotherapy, biologic, or hormonal therapy for cancer treatment used concurrently or within 6 months prior to first dose of study treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
18. Major surgery (as defined by the Investigator) within 4 weeks prior to starting the study; patients must have recovered from effects of preceding major surgery. Note: Local non-major surgery for palliative intent (e.g., surgery of isolated lesions) is acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS1) | 2 years
  Progression Free Survival using investigator assessments according to Response Evaluation Criteria in Solid Tumours (RECIST 1.1) defined as number of months from first dose of chemotherapy until last follow-up, PD, death or withdrawal of consent.

SECONDARY OUTCOMES:
Progression Free Survival (PFS0) | for a minimum of 24 months from inclusion
  Progression Free Survival using investigator assessments according to Response Evaluation Criteria in Solid Tumours (RECIST 1.1) defined as number of months from first dose of osimertinib until last follow-up, PD, death or withdrawal of consent.
Overall Survival (OS1) | for a minimum of 24 months from inclusion
  OS1 Survival will be calculated from the first dose of chemotherapy until the date of death from any cause. If no event is observed (e.g. lost to follow-up) OS is censored at the day of last subject contact.
Overall Survival (OS0) | for a minimum of 24 months from inclusion
  OS0 Survival will be calculated from the date of start of osimertinib until the date of death from any cause. If no event is observed (e.g. lost to follow-up) OS is censored at the day of last subject contact.
Incidence of treatment related Adverse Events (Safety and Tolerability) | up to 16 weeks from start of study treatment
  Frequency and severity of Adverse Events, grading according to CTCAE V5.0
Measurement of Quality of Life with PRO-CTCAE. questionnaire | up to 16 weeks from start of study treatment
  Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) minimum value: not at all (1); maximum value: severe (5); higher scores mean a worse outcome
Measurement of Quality of Life with EORTC QLQ-C30 questionnaire | up to 16 weeks from start of study treatment
  The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) minimum value: not at all (1); maximum value: very much (4); higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sebastian, MD, Principal Investigator — Goethe University Frankfurt
Locations (16):
- Germany (16):
  - Charité Universitätsmedizin Berlin Campus Virchow Klinikum Klinik mit Schwerpunkt Infektiologie und Pneumologie, Berlin
  - Universitätsklinik Köln, Lung Cancer Group Cologne - Innere Medizin I, Cologne
  - Technische Universität Dresden Medizinische Fakultät Carl Gustav Carus Medizinische Klinik und Poliklinik I, Dresden
  - Universitätsklinikum Essen, Westdeutsches Tumorzentrum - Innere Klinik, Essen
  - University Hospital Frankfurt, Frankfurt
  - Asklepios Lungenklinik Gauting, Gauting
  - MVZ II der Niels Stensen Kliniken; Franziskus Hospital Harderberg, Georgsmarienhütte
  - Universitätsmedizin Göttingen, Klinik für Hämatologie und Medizinische Onkologie, Göttingen
  - Krankenhaus Martha-Maria Halle-Dölau Klinik für Innere Medizin II, Halle
  - Universitätsklinikum Hamburg-Eppendorf Hubertus Wald Tumorzentrum - UCCH II. Medizinische Klinik und Poliklinik, Hamburg
  - Universitätsklinikum Heidelberg, Thoraxklinik Heidelberg gGmbH, Heidelberg
  - DGD Lungenklinik Hemer, Hemer
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - LMU-München Pneumologie und Thorakale Onkologie Medizinische Klinik V; Innenstadt, München
  - Klinikum Nürnberg Nord Paracelsus Med. Privat Universität Pneumologie und Lungentumorzentrum, Nuremberg
  - Pius Hospital Oldenburg Medizinischer Campus Universität Oldenburg, Oldenburg

IPD SHARING:
Plan to Share IPD: No